CLINICAL TRIAL: NCT07181759
Title: Prospective Randomized Controlled Clinical Trial on the Treatment of Upper Urinary Tract Stones With VISOR and fURS
Brief Title: Clinical Trial of VISOR vs fURS for Upper Urinary Tract Stone
Acronym: VISOR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-R042-02
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Urolithiasis, Calcium Oxalate; Ureteroscopy; Therapeutic Irrigation; Intraoperative Complications
Keywords: Ureterorenoscopy; Upper urinary tract calculi; Intrarenal pressure; Stone-free rate (SFR); Lithotripsy; VISOR; Vortex intelligence Stone Optimized Removal(VISOR）
MeSH Terms: conditions — Nephrolithiasis, Calcium Oxalate; Intraoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VISOR (Experimental): Surgery will be performed using the VISOR through a 14Fr UAS
  Interventions: Procedure: VISOR
- fURS (Active Comparator): Surgery will be performed using a standard single-use electronic ureterorenoscope through a 14Fr UAS
  Interventions: Procedure: fURS

INTERVENTIONS:
Procedure: VISOR — Surgery will be performed using the VISOR through a 14Fr UAS
  Arms: VISOR
Procedure: fURS — Surgery will be performed using a standard single-use electronic ureterorenoscope through a 14Fr UAS
  Arms: fURS

SUMMARY:
This prospective randomized controlled clinical study aims to evaluate the safety and efficacy of a novel Vortex Intelligence Stone Optimized Removal (VISOR,The experimental group) system compared to a single-use ureterorenoscope (the control) for treating upper urinary tract stones.

A total of 100 patients with upper urinary tract stones (cumulative stone diameter ≤3 cm) will be enrolled and randomly assigned in a 1:1 ratio to either the experimental group (n=50) or the control group (n=50). The experimental group will undergo surgery using the innovative system, which integrates irrigation-suction, pressure monitoring-regulation, and lithotripsy-evacuation functions. The control group will be treated with a conventional single-use ureterorenoscope.

The primary outcome measure is the immediate stone-free rate (SFR), defined as the proportion of patients with residual fragments <4 mm on renal non-contrast computed tomography (NCCT) performed within 24 hours postoperatively. Key secondary endpoints include the SFR at 3 months, operative and lithotripsy times, total laser energy used, intraoperative ureteral injury (Traxer grading), postoperative pain scores, incidence of fever (>38.0°C), and overall complication rates (Clavien-Dindo classification).

Patient follow-up assessments will be conducted at 24 hours, 21±7 days, and 90±14 days post-surgery to monitor stone clearance, complications, and recovery. This study seeks to determine if the novel system offers superior stone clearance while maintaining a safe renal pelvic pressure profile, potentially improving outcomes for patients with larger renal stones treated ureteroscopically.

DETAILED DESCRIPTION:
1. Study Background and Rationale

   Urolithiasis is a highly prevalent urological disease, ranking first among inpatient admissions in urology departments. It is characterized by high incidence and recurrence rates. In China, the incidence ranges from 1% to 5%, with higher rates in the eastern and southern regions, reaching 5-10% in the south. Approximately 150-200 new cases per 100,000 people require hospitalization each year, with a rising trend establishing China as one of the world's three high-risk regions for stones.

   The primary surgical treatments for renal stones are flexible ureteroscopy (fURS) and percutaneous nephrolithotomy (PCNL). fURS, utilizing the natural urinary tract, is minimally invasive with fewer complications but is limited by lower lithotripsy efficiency, making it guideline-recommended for stones <2cm. PCNL, while highly efficient for stones >2cm, carries higher risks, including significant bleeding and potential injury to adjacent organs.

   There is a growing trend to use fURS for larger stones (>2cm), yet several challenges remain:

   Low Lithotripsy Efficiency: Small working channels limit laser fiber size, requiring dusting, which clouds the visual field.

   Difficulty in Stone Retrieval: Incomplete clearance, especially in the lower pole, leads to residual fragments, increasing the risk of obstruction and recurrence.

   Uncontrolled Intrarenal Pressure (IRP): Obstruction of the ureteral access sheath (UAS) can cause elevated IRP, leading to fluid absorption and life-threatening urosepsis. Current suction techniques are inefficient at pressure control.

   Multiple Procedures: The above issues often necessitate multiple surgeries, increasing patient burden.

   While technological advances like high-power lasers and the "dusting" technique have expanded fURS applications, the fundamental problems of fragment clearance and IRP control persist. The novel Vortex Intelligence Stone Optimized Removal System(VIROS) is designed to address these limitations by integrating irrigation-suction, pressure monitoring-regulation, and lithotripsy-evacuation into a single platform. This study aims to rigorously evaluate whether this system can improve stone-free rates while maintaining a safer intraoperative pressure profile compared to standard single-use fURS.
2. Study Objectives

   Primary Objective: To compare the postoperative immediate stone-free rate (SFR) at 24 hours between the experimental system and the single-use fURS.

   Secondary Objectives: To compare the two groups regarding:

   SFR at 3 months postoperatively. Intraoperative parameters (ureteroscopy operation time, lithotripsy time, total laser energy).

   Safety outcomes (Traxer ureteral injury grade, postoperative complications per Clavien-Dindo classification, postoperative fever rate).

   Postoperative pain scores (VAS).
3. Study Design

   Design: Prospective, randomized, controlled, single-blind (outcome assessor), parallel-group clinical trial.

   Sample Size: 100 participants. Randomization: 1:1 allocation to experimental or control group using a computer-generated randomization schedule. Opaque sealed envelopes will be used to conceal allocation until intervention.

   Blinding: Due to the nature of the devices, surgeons and patients cannot be blinded. However, radiologists assessing the primary outcome (CT scans for stone clearance) and data analysts will be blinded to group assignment.
4. Study Population

   Inclusion Criteria: Adults (≥18 years) with upper urinary tract stones (cumulative diameter ≤3cm) scheduled for fURS holmium laser lithotripsy, who can provide informed consent.

   Exclusion Criteria: Key exclusions include need for bilateral surgery, significant hydronephrosis (≥4cm), previous renal/ureteral surgery, active infection/fever, pregnancy, severe comorbidities (ASA≥3), renal anatomical anomalies, coagulation disorders, and concurrent participation in another trial.
5. Interventions

   Experimental Group: Surgery will be performed using the Vortex-Assisted Stone Removal Ureterorenoscopy System (Double-channel pressure-measuring electronic ureterorenoscope, Model: XY-MU-12-620S) through a 14Fr UAS. The system's integrated suction and pressure monitoring functions will be utilized throughout the procedure.

   Control Group: Surgery will be performed using a standard single-use electronic ureterorenoscope (Model: XY-S650A) through a 14Fr UAS, following conventional surgical protocols without the integrated suction/pressure control of the experimental system.

   All other surgical, anesthetic, and perioperative care protocols will be identical for both groups.
6. Study Procedures and Timeline

   Screening (Day -14 to 0): Informed consent, eligibility assessment, collection of baseline demographics and medical history, and pre-operative tests (lab tests, ECG, NCCT).

   Treatment (Day 0): Randomized surgery. Intraoperative data (times, laser energy, Traxer grade) and adverse events are recorded.

   Post-op 24 Hours: Pain assessment (VAS), temperature monitoring, complication assessment, and NCCT to evaluate the primary outcome (immediate SFR). Blood tests (CRP, IL-6, PCT) are repeated to monitor for infection.

   Follow-up 1 (21 ± 7 days): Clinical review, decision on stent removal based on post-op Day 1 CT findings, recording of adverse events and unplanned readmissions.

   Follow-up 2 (90 ± 14 days): Final NCCT to determine secondary outcome (3-month SFR), assessment of hydronephrosis, and recording of any late adverse events or re-interventions.
7. Outcome Measures

   Primary Endpoint: Immediate Stone-Free Rate (SFR), defined as the absence of residual fragments ≥4mm on NCCT within 24 hours post-surgery.

   Secondary Endpoints:

   SFR at 90 days (residual fragments <4mm). Ureteroscopic operation time (from scope entry to exit). Total lithotripsy time and total laser energy (Joules). Intraoperative ureteral injury (Traxer grading scale, 0-4). Postoperative pain (Visual Analog Scale, 0-10). Incidence of postoperative fever (body temperature ≥38.0°C). Postoperative complication rate and severity (Clavien-Dindo Classification).
8. Data Analysis

Statistical analyses will be performed using appropriate software (e.g., SPSS, R). The difference in the primary outcome (immediate SFR) between groups will be analyzed using Chi-square or Fisher's exact test. Continuous variables (e.g., operation time, pain scores) will be compared using Student's t-tests or Mann-Whitney U tests depending on data distribution. A p-value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper urinary tract stones and a cumulative stone diameter ≤3 cm;
* Patients scheduled to undergo "flexible ureteroscopic holmium laser lithotripsy";
* Age ≥18 years;
* Patients without psychiatric disorders or language dysfunction, capable of understanding the study and providing informed consent.

Exclusion Criteria:

* Patients requiring bilateral lithotripsy in a single-stage ureteroscopic procedure;
* Ipsilateral hydronephrosis with >4 cm renal pelvic separation;
* Patients with a history of open or laparoscopic renal and/or ureteral surgery;
* Fever (body temperature ≥38°C) due to urinary tract infection or other causes within one week prior to surgery;
* Pregnant women;
* Patients with severe systemic diseases, cardiac diseases, pulmonary insufficiency, or vital organ failure unable to tolerate anesthesia or surgery (ASA score ≥3);
* Patients with anatomical abnormalities such as polycystic kidney, horseshoe kidney, or ectopic kidney;
* Patients with coagulation disorders (e.g., INR >2.0 or platelet count <80×10⁹/L);
* Patients currently participating in other device or drug clinical trials;
* Patients deemed ineligible for the trial by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Immediate Postoperative Stone-Free Rate (SFR): | 24 hours after surgery
  Stone clearance rate within 24 hours after surgery.

SECONDARY OUTCOMES:
Stone-Free Rate at 3 Months Postoperatively | 3 Months Postoperatively
  Stone-Free Rate at 3 Months Postoperatively

OTHER OUTCOMES:
Ureteroscopy Operation Time: | Juring Operation
  Duration from the insertion of the flexible ureteroscope to its removal.
Lithotripsy Time | Juring operation
  Time spent on lithotripsy
Total Laser Energy | Juring operation
  Total laser energy delivered (in joules)
Traxer Ureteral Injury Grading | Juring Operation
  Grade 0: No injury or only mucosal bleeding. Grade 1: Ureteral mucosal injury without involvement of the smooth muscle layer.
  Grade 2: Ureteral wall injury involving the mucosa and smooth muscle layers, without penetration of the adventitia (no visible fat tissue).
  Grade 3: Ureteral wall injury involving the mucosa and smooth muscle layers, with penetration of the adventitia (fat tissue visible).
  Grade 4: Complete ureteral tear.
Postoperative Pain Score | Within 24 hours after surgery
  Assessed using the Visual Analog Scale (VAS), where 0 indicates no pain and 10 indicates the worst pain imaginable
Postoperative Fever | 72 hours After Operation
  Rate of participant temperature exceeding 38.0°C after surgery.
Postoperative Clavien-Dindo Classification of Surgical Complications. | 72 hours After Operation
  Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventionsAllowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
  Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.Blood transfusionsand total parenteral nutritionare also included.
  Grade III Requiring surgical, endoscopic or radiological intervention- IIIa；Intervention not under general anesthesia - IIIb
  Intervention under general anesthesia-Grade IV
  Grade V Death of a patient
  Life-threatening complication (including CNS complications)* requiring IC/ICU-management- IVa；single organ dysfunction (including dialysis) - IVb multiorgan dysfunction

IPD SHARING:
Plan to Share IPD: No